CLINICAL TRIAL: NCT03713450
Title: A Prospective Single Centre Randomized Interventional Controlled Trial Comparing Patient and Staff Safety During Aorto-iliac Revascularization Procedures Under Automated Fusion Imaging Guidance With Controls
Brief Title: Patient and Staff Safety During Aorto-iliac Revascularization Procedures Under Automated Fusion Imaging Guidance With Controls
Acronym: CYDAR ILIAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Premature termination of the research following an internal reorganization of the team no longer allowing the necessary resources to continue the study
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC18_0092
Record Dates: First submitted 2018-10-18; First posted 2018-10-19 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Patient and Staff Radiation Exposure During Aorto-iliac Endovascular Revascularization
Keywords: Radiation; Contrast; Endovascular; Fusion imaging guidance; Iliac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control with imaging guidance (Experimental)
  Interventions: Device: Control with imaging guidance
- Control without imaging guidance (Active Comparator)
  Interventions: Device: Control without imaging guidance

INTERVENTIONS:
Device: Control with imaging guidance — Prospective randomized study during aorto-iliac revascularisation comparing patient and staff radiation exposure using the automated overlay imaging guidance, in addition to the application of the ALARA principles.
  The study includes only the per-operative period but no follow-up. The study will be performed in all imaging environment (Hybrid room or mobile).
  Arms: Control with imaging guidance
Device: Control without imaging guidance — Prospective randomized study during aorto-iliac revascularisation comparing patient and staff radiation exposure not using the automated overlay imaging guidance, in addition to the application of the ALARA principles.
  The study includes only the per-operative period but no follow-up. The study will be performed in all imaging environment (Hybrid room or mobile).
  Arms: Control without imaging guidance

SUMMARY:
Endovascular revascularization has revolutionized the field of vascular surgery and has become the first-choice treatment for peripheral arteries occlusive disease. However, the drawback of this technic is the X-ray exposure for both patients and staff and the iodinated contrast injection for the patient.

One way to reduce both radiation and contrast use is to use advanced imaging techniques allowing an overlay of a 3D vascular mask (from a pre-operative CT scan) onto the live X-ray image. This has been proven during endovascular aneurysm repair.

This advanced imaging application is currently available only in the latest expensive hybrid operating rooms, requires additional manoeuvre from the operator throughout the procedure, and may be X-rays and contrast consuming.

This trial will examine the clinical benefits based on patient and staff' radiation exposure during aorto-iliac revascularisation, of a new software imaging guidance, suitable for any theatre including those equipped with mobile C-arm, fully automated and with a radiation free overlay registration process.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 or older,
* Patients scheduled for aorto iliac endovascular revascularisation,
* Pre-operative CT scan.

Exclusion Criteria:

* Women of childbearing age,
* Absence of preoperative CT scan,
* Emergency procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Dose area product | The end of the procedure
  Dose area product (DAP) by the end of the procedure.

SECONDARY OUTCOMES:
Number of DSA runs | The end of the procedure
  Number of DSA runs by the end of the procedure.
Air Kerma | The end of the procedure
  Air Kerma (mGy) by the end of the procedure.
Fluoroscopy time | The end of the procedure
  Fluoroscopy time (min) by the end of the procedure.
Contrast volume | The end of the procedure
  Contrast volume (ml) by the end of the procedure.
Operative time | The end of the procedure
  Operative time (min) by the end of the procedure.
Operator exposure | The end of the procedure
  Operator exposure (Sv) by the end of the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Vascular surgery, Institut du Thorax, Nantes, France

IPD SHARING:
Plan to Share IPD: No